CLINICAL TRIAL: NCT04959149
Title: A Comparison of Face-to-face Endotracheal Intubation and Typical Intubation With Airtraq Video Laryngoscope in Bariatric Patients: a Randomised Controlled Trail
Brief Title: Face-to-face Intubation in Morbidly Obese
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Lodz (Other)
Responsible Party: Principal Investigator, Tomasz Gaszynski, professor of anaesthesia, Medical University of Lodz
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: RNN/62/20/KE
Record Dates: First submitted 2020-12-28; First posted 2021-07-13 (Actual); Last update posted 2022-06-10 (Actual); Status verified 2022-06

CONDITIONS: Intubation;Difficult; Obesity, Morbid
Keywords: obesity; intubation; videolaryngoscope
MeSH Terms: conditions — Obesity, Morbid; Obesity

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- face-to-face intubation (Experimental): intubation approach from front of the patient
  Interventions: Device: AirTraq videolaryngoscope
- standard position intubation (Active Comparator): intubation approach from behind the head of the patient
  Interventions: Device: AirTraq videolaryngoscope

INTERVENTIONS:
Device: AirTraq videolaryngoscope — intubation of morbidly obese patient using Airtraq videolaryngoscope

SUMMARY:
Introduction : In a typical endotracheal intubation, the patient is in the supine position, with the anesthetist standing behind his head and with adequate access to the head and neck of the patient. However, there are several situations, where traditional intubation is very difficult or even impossible. In immobilised trauma victims, with limited access to the head, suspected cervical spine injury or in sitting positioned patient an intubation performed by a person standing in front of a patient might be the only chance of airway management. Moreover, in case of general anesthesia in bariatric patients, face-to-face (inverse) method is increasingly being considered due to upper body elevation position, recommended in this group of patients.

This was a parallel randomised controlled trial in patients scheduled for planned sleeve gastrectomy in Barlicki University Hospital, Lodz, Poland. Randomization and allocation to trial group were carried out by drawing envelopes by independent observer before a procedure. Randomized and recruited participants were 76 adults (typical intubation n= 36, face-to-face intubation n=40). Main outcome was a time of intubation using Airtraq video laryngoscope measured by independent assistant.

DETAILED DESCRIPTION:
Aim : The aim of the study is to evaluate the effectiveness and safety of face-to-face intubation in airway management.

Methods : Patients admitted to hospital for elective sleeve gastrectomy procedure will be included in the study protocol. Before induction of anaesthesia the draw of the method will be held. The choice of method of intubation (inverse or typical) will be random.

1. All patients will be positioned with the elevation of the upper body about 30 degrees. The standard anesthesia monitoring involves electrocardiogram, pulsoxymetry, non-invasive blood pressure and end-tidal carbon dioxide.
2. Patients will be pre-oxygenated for 5 min. with 100% oxygen using facemask.
3. The induction of general anesthesia will be performed by the intravenous administration of 1-2 µg.kg-1 of fentanyl and 2-2,5 mg.kg-1 propofol.
4. After mask ventilation possibility is confirmed, rocuronium in a dose of 0,6 mg.kg-1 will be given.
5. After obtaining an optimal muscle relaxation (90 s.) patient will be intubated. In face-to-face method an anesthetist is standing in front of a patient. In typical intubation an anesthetist is standing behind the patient's head.
6. In case of prolonged face-to-face intubation (>120 s) or 2 unsuccessful attempts, patients are supposed to be intubated in a traditional way with the same video laryngoscope.
7. General anesthesia will be continued with desflurane and a mixture of the oxygen and air, volume-controlled ventilation parameters will be adjusted to age and ideal body weight.

ELIGIBILITY:
Inclusion Criteria:

1. BMI > 40 kg.m-2
2. Patients qualified for planned sleeve gastrectomy.
3. Patients of I and II class of ASA scale.
4. Patients without history of difficult intubation.

Exclusion Criteria:

1. Patients in life threatening states.
2. Patients of III, IV, V and VI class of ASA scale.
3. History of difficult intubation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Actual)
Dates: Start 2020-03-01 (Actual); Primary Completion 2020-09-01 (Actual); Study Completion 2020-09-30 (Actual)

PRIMARY OUTCOMES:
time of intubation | during the intervention/procedure
  time of intubation measured from grabbing the device to confirming the correct placement using EtCO2

SECONDARY OUTCOMES:
effectiveness | during the intervention/procedure
  effectiveness as number of correct placement of endotracheal tube in the trachea of the patient

OTHER OUTCOMES:
complications | immediately after the intervention/procedure
  complications defined as soft tissue injuries ex lips or mucosa of oral cavity injury, sore throat after extubation, desaturations below 92%

CONTACTS AND LOCATIONS:
Overall Officials: Tomasz Gaszynski, Principal Investigator — Medical University of Lodz, Poland
Locations (1):
- Medical University of Lodz, Poland, Lodz, Poland

IPD SHARING:
Plan to Share IPD: No
on request

REFERENCES:
- [Background] Arslan ZI, Alparslan V, Ozdal P, Toker K, Solak M. Face-to-face tracheal intubation in adult patients: a comparison of the Airtraq, Glidescope and Fastrach devices. J Anesth. 2015 Dec;29(6):893-8. doi: 10.1007/s00540-015-2052-6. Epub 2015 Jul 29. PMID 26219732
- [Background] Jeong H, Chae M, Seo H, Yi JW, Kang JM, Lee BJ. Face-to-face intubation using a lightwand in a patient with severe thoracolumbar kyphosis: a case report. BMC Anesthesiol. 2018 Jul 21;18(1):92. doi: 10.1186/s12871-018-0556-y. PMID 30031381